CLINICAL TRIAL: NCT01496898
Title: Vaginal Microflora and Inflammatory Markers Before and After Levonorgestrel Device Insertion
Brief Title: Changes in Vaginal, Cervical and Uterine Microflora With Levonorgestrel Intrauterine Device Placement
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: uufpf 43416
Record Dates: First submitted 2011-08-21; First posted 2011-12-21 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Human Microbiome; Metagenome; Contraception; Cytokine
Keywords: Microflora; Vaginal; Cervical; Uterine; Inflammation; Cytokine; Intrauterine Device; Levonorgestrel
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A total of 648 samples will be collected from 12 participants for bacterial species and human cytokine analysis in 9 collection visits. Specimens will be collected up to one week prior to IUD insertion and two months after IUD insertion. Vaginal and cervical specimens will be collected using FLOQSwabs® (Copan) to maximize bacterial DNA sample collection. Uterine samples will be collected by uterine irrigation with sterile saline using an embryo replacement catheter.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this study is to examine changes in the bacterial ecology and inflammatory markers of the female genital tract with levonorgestrel intrauterine device placement.

The specific research objectives of this project include:

1. Characterization of vaginal, cervical and uterine bacterial species and communities prior to and after LNG IUD placement using bacterial DNA microarray analysis. Samples will be collected up to 1 week before and 2 months after IUD insertion.
2. Characterization of vaginal, cervical and uterine inflammatory cytokine milieu prior to and after LNG IUD placement using human RNA microarray analysis. Samples will be analyzed from up to one day before and three weeks after IUD insertion.
3. Establish a tissue bank of vaginal, cervical and uterine specimens for future research.

ELIGIBILITY:
Inclusion Criteria:

* Not currently pregnant
* No use of hormonal birth control for at least three months prior to enrollment
* Desiring levonorgestrel IUD for birth control
* Greater than 6 months postpartum
* Greater than 6 weeks after miscarriage
* No antibiotic use in the past 6 weeks

Exclusion Criteria:

* Uterine Abnormalities
* Current use of hormonal contraceptives or use less than 3 months ago
* Unexplained vaginal bleeding
* Irregular menses
* Cervical dysplasia
* Cervical or vaginal infection in the last 6 weeks
* Douching within the week prior to sample collection
* Use of vaginal lubricants within the week prior to sample collection

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Caucasian woman aged 18 to 45 seeking intrauterine contraception meeting inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Changes in vaginal, cervical and uterine bacterial species with levonorgestrel intrauterine device placement | 1 week prior to IUD insertion to 2 months after IUD insertion
  Characterization of vaginal, cervical and uterine bacterial species and communities prior to and after LNG IUD placement using bacterial DNA microarray analysis

SECONDARY OUTCOMES:
Inflammatory cytokine changes with levonorgestrel intrauterine device placement | 1 day prior to IUD insertion to 3 weeks after IUD insertion
  Characterization of vaginal, cervical and uterine inflammatory cytokine milieu prior to and after LNG IUD placement using human RNA microarray analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Janet C Jacobson, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Hospital, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Jacobson JC, Turok DK, Dermish AI, Nygaard IE, Settles ML. Vaginal microbiome changes with levonorgestrel intrauterine system placement. Contraception. 2014 Aug;90(2):130-5. doi: 10.1016/j.contraception.2014.04.006. Epub 2014 Apr 21. PMID 24835828